CLINICAL TRIAL: NCT01514344
Title: Phase II Study on Activity and Tolerability of Intralesional Rituximab in Patients With Relapsed or Refractory CD20+ Indolent Lymphomas of Conjunctiva; Activity of Supplemental Autologous Serum in Patients Not Responsive to Rituximab Alone
Brief Title: Intralesional Rituximab for the Treatment of Conjunctival Indolent Lymphoma
Acronym: IRIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andres J. M. Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andres J. M. Ferreri, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRIS
Record Dates: First submitted 2012-01-06; First posted 2012-01-23 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Ocular Adnexal Mucosa-Associated Lymphoid Tissue Lymphoma
Keywords: OAL; MALT; conjunctiva; indolent; CD20+
MeSH Terms: interventions — Rituximab; Complement System Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intralesional rituximab (Experimental)
  Interventions: Drug: intralesional rituximab; Biological: supplemental autologous serum

INTERVENTIONS:
Drug: intralesional rituximab — 10-20 mg (1-2 ml) rituximab once a week for 4 weeks; followed by 10-20 mg (1-2 ml) rituximab monthly per six months
  Other Names: Intraconjunctival rituximab; mabthera, anti-CD20 therapy
Biological: supplemental autologous serum — patients in PD or SD during or after administration of 6 doses monthly rituximab will be administered the same dose of intralesional rituximab supplemented by autologous serum
  Other Names: autologous serum supplementation; complement

SUMMARY:
Phase II, monocentric, open label study to assess safety and activity of intralesional Rituximab for the treatment of indolent CD20+ lymphoma of conjunctiva.

DETAILED DESCRIPTION:
Preliminary data suggest intralesional rituximab is able to revert resistance to systemic rituximab in patients with CD20+ indolent lymphoma of the conjunctiva, and the addition of autologous serum seems to exhibit a synergistic effect on tumor regression. These two main aspects will be assessed in this trial.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of CD20+ B cell lymphoma subtypes: marginal zone lymphoma, grade 1-2 follicular lymphoma, plasmocytic lymphoma, small lymphocyte lymphoma
* conjunctival localization alone (1EA stage; mono- or bilateral)
* at least one measurable lesion
* age >/= 18 years
* ECOG-PS </=3
* HIV 1-2 negativity
* at least one previous treatment (antibiotic or rituximab)

Exclusion Criteria:

* concomitant conventional (chemo-, radiation, immuno-), experimental (antibiotic) or corticosteroid anticancer therapy
* known allergy to rituximab
* systemic symptoms
* concurrent diagnosis of pemphigus
* postsurgical conjunctival scars

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
assessment of safety | During experimental treatment (within 7 months from trial registration)
  assessment of safety of intralesional rituximab in terms of incidence of >/= G4 adverse events during the experimental treatment

SECONDARY OUTCOMES:
assessment of activity | at the end of experimental treatment (at 7th month from trial registration)
  assessment of activity of intralesional rituximab in terms of overall partial and complete response and duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — San Raffaele Scientific Institute, Milano, Italy
Locations (1):
- Dip. Oncoematologia - Fondazione Centro San Raffaele del Monte Tabor, Milan, Italy

REFERENCES:
- [Derived] Ferreri AJM, Sassone M, Miserocchi E, Govi S, Cecchetti C, Corti ME, Mappa S, Arcaini L, Zaja F, Todeschini G, Mannina D, Calimeri T, Perrone S, Ponzoni M, Modorati G. Treatment of MALT lymphoma of the conjunctiva with intralesional rituximab supplemented with autologous serum. Blood Adv. 2020 Mar 24;4(6):1013-1019. doi: 10.1182/bloodadvances.2020001459. PMID 32182364